CLINICAL TRIAL: NCT03704922
Title: Age of Blood in Sickle Cell Transfusion -The Effects of Phosphotidylserine Expression on Older Red Cell Units in Adults With Sickle Cell Disease
Brief Title: Age of Blood in Sickle Cell Transfusion
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-0018; K23HL136787-01 (NIH)
Record Dates: First submitted 2018-10-05; First posted 2018-10-15 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-07

CONDITIONS: Sickle Cell Disease
Keywords: Transfusion
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ≤10 day Blood (Experimental): Subjects in this group will receive only blood stored ≤10 days for 3 consecutive transfusion events.
  Interventions: Biological: Transfusion
- ≥30 day Blood (Experimental): Subjects in this group will receive only blood stored ≥30 days for 3 consecutive transfusion events.
  Interventions: Biological: Transfusion

INTERVENTIONS:
Biological: Transfusion — Red cell units for transfusion

SUMMARY:
The Investigators hypothesize that older red cell units trigger phagocytosis and activation of circulating macrophages with a downstream immunomodulatory cascade and release of excess Non Transferrin Bound Iron(NTBI) that leads to increased rates of infection in adults with Sickle Cell Disease(SCD).

To test this hypothesis, the study staff will perform a randomized prospective clinical trial. In aim 1, the study staff will determine the biochemical differences between ≥30 day-old versus ≤10 day-old units. In aim 2, the study staff will determine the physiologic effects of the transfused blood in a patient with SCD. Lastly, in aim 3, the study staff will explore the clinical implications of receiving older red cells over a 3 month period.

DETAILED DESCRIPTION:
The Investigators assembled a multidisciplinary investigative team to examine the potential effects of older red cell units in adults with Sickle Cell Disease(SCD). Study staff have preliminary data that show: 1) there is equipoise among blood bank directors about the effects of older units in adults with SCD, 2) in our institution, many adults are administered older units, 3) older units activate macrophages and 4) this physiology promoted by older units is associated with an increased risk of infection. Our team is now poised to take the next investigative step: a prospective, randomized study.

In Milwaukee, 1/3 of units transfused to adults with SCD are >30 days old, but nation-wide some restrict the transfusion of older units. About four hundred adults receive care in the Adult Sickle Cell Clinic at Froedtert Hospital in Milwaukee, about 23 of who receive chronic outpatient transfusions for chronic pain or stroke prophylaxis. Transfusions are administered to adults regardless of storage age, except in the case of red cell exchange, for which there is a policy to use less than 14 day old units. In a 3-year retrospective review of transfusions administered to adults with SCD, 627 units were given via simple transfusion over 281 outpatient encounters. The overall median unit storage age was 22 days (range: 2-42 days), and 25% of the units transfused were stored 33 days or longer.

To determine the opinions and policies of other hospital blood bank directors about the use of older red cell units for patients with SCD, study staff conducted a nation-wide survey (n=90). While only 23% of respondents had a storage age restriction policy for patients with SCD, 31% thought that older units were not as effective as younger units, and 65% believed that evidence-based policies were needed

Adults with SCD may be susceptible to the effects of an older unit's physiology because they are prone to infection, inflamed, and poorly equipped to handle excess iron. In a cohort of 40 steady-state adults with SCD, the investigators specifically measured markers of inflammation and iron excess. High sensitivity C-reactive protein, a marker of systemic inflammation, was found to be markedly elevated (median 5.6 mg/L, range 0.4-60 mg/L; reference range <1.0 mg/L), as was ferritin, a marker of iron stores (median 2,969 ng/ml, range 20-12,300 ng/ml; reference range 13-400 ng/ml).

Forty chronically-transfused adults with SCD will be randomized in a double-blind fashion to receive ≥30 day-old or ≤10 day-old units for, at most, 3 consecutive outpatient transfusions. Subjects will be randomized in blocks of 5 and stratified by age: at least 10 subjects from each of the age ranges 16-30 and 31-60 years will be enrolled. Pre-transfusion, sterile samples will be extracted from red cell units. Patient peripheral blood will be also obtained 1 month before randomization, immediately pre-transfusion, and 2 and 24 hours post-transfusion. Hemoglobin will be measured pre-transfusion, 2 and 24 hours post-transfusion, and 2 weeks post transfusion. Participants will complete standardized diaries daily to document symptoms of infection, SCD pain, medications and Emergency Department(ED) or hospital use. Diaries will be collected and participants will be assessed with each transfusion encounter and 4 weeks after the last transfusion. To ensure compliance, coordinators will contact subjects weekly to complete the diaries.

Study staff will evaluate red cells pre- and post-transfusion for Phosphatidylserine(PE), Phosphatidylethanolamine (PS), and microparticles as above for all blood samples. White cells will be isolated with established separation techniques. The white cell populations of interest will be defined by their location on a forward scatter/side scatter plot and their positivity using key fluorochrome-labeled identity markers (macrophages: CD14, neutrophils: CD16). Once the cell populations of interest are identified, the cells will be evaluated for various markers of activation. The plasma fraction from each patient and red cell unit will be diverted to determine concentrations of free heme/hemoglobin, cytokines, and NTBI, respectively.

ELIGIBILITY:
Inclusion Criteria:

* age 16 to 60 years
* have diagnosis of sickle cell disease
* receiving outpatient red cell transfusion therapy
* outpatient at the time of transfusion

Exclusion criteria:

* history of reactions to transfusion therapy that cannot be adequately managed by antihistamines
* do not have crossmatch compatible red cells
* participation in another therapeutic trial for SCD
* pregnant
* HIV positive
* uncontrolled inter-current illness, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Little, MD, Principal Investigator — University of North Carolina, Chapel Hill; Matthew Karafin, MD, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Versiti Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 to 36 months following publication
Access Criteria: IRB, IEC, or REB approval and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Karafin MS, Fasano RM, Ilich A, Wichlan D, Chang A, Janecke R, Zellner-Jones S, James SM, Butler HE, Kolupaev O, Caughey MC, Wilson SR, Key NS, Field JJ, Little JA. Red cell physiologic stress results in lower quality transfusions: a randomized trial in adults with sickle cell disease. Blood Red Cells Iron. 2025 Dec;1(3):100017. doi: 10.1016/j.brci.2025.100017. Epub 2025 Oct 1. PMID 41312340
- [Derived] Karafin MS, Grier AL, Fasano RM, Ilich A, Wichlan D, Chang A, James SM, Butler HE, Kolupaev O, Caughey MC, Stephenson DJ, Reisz JA, Key NS, Field JJ, Little JA, Spitalnik SL, D'Alessandro A. Blood-storage duration affects hematological and metabolic profiles in patients with sickle cell disease receiving transfusions. J Clin Invest. 2025 Jul 3;135(17):e192920. doi: 10.1172/JCI192920. eCollection 2025 Sep 2. PMID 40608427

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ≤10 Day Blood | ≥30 Day Blood
Started | 13 | 13
Completed | 10 | 10
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ≤10 Day Blood | ≥30 Day Blood | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (8.5) | 29.8 (11.2) | 30.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 13 | 26
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Biochemically Old Red Cell Units
Description: The investigators will compare the transfusions provided to the two groups (the proportion of biochemically old units when stored ≥30 days compared to when stored ≤10 days) using a Fisher exact test at an alpha of 0.05.
Time Frame: through third transfusion, an average of 18 weeks
Measure: Number; unit: proportion biologically old units
Arm/Group | ≤10 Day Blood | ≥30 Day Blood
Number analyzed (Participants) | 13 | 13
proportion biologically old units | 0.71 | 0.86
Statistical Analysis 1: Comparison: ≤10 Day Blood vs ≥30 Day Blood; Test type: Other; p = 0.051, Fisher Exact

2. Other Pre Specified Outcome: Change in the Concentration of CD62L Positive Circulating Monocytes
Description: Change in CD62Lcirculating monocyte/macrophage mean fluorescence intensity (MFI) at 2 hours post-transfusion compared to the subject pre-transfusion. The investigators will compare the two groups using a two sample two-sided t-test of the log at an alpha of 0.05. Power: In addition, we will use a generalized linear model to include biochemically old units transfused,regardless of unit age, as a covariate. Other co-variates will include free heme, cell free hemoglobin, and non-transferrin bound iron (NTBI) from the transfused unit. We will similarly compare secondary activation endpoints: activation markers for neutrophils and measured cytokine concentrations. When possible, donor and recipient red cells will be differentiated in S-antigen negative patients who are by chance provided S-positive heterozygous or homozygous donor red cells.
Time Frame: through third transfusion, an average of 18 weeks
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Percentage of Infections in Adults
Description: The primary endpoint is the percentage of infections in adults who receive ≥30 day-old units as compared to ≤10 day-old units. The presence of an indwelling catheter will be used as a key co-variate in this analysis.
  The investigators will further explore the relationship of blood age and transfusion of biochemically old red cell units on the change in hemoglobin (Hb) and hemoglobin S (HbS)% over time, daily pain scores, opioid use and dose, emergency department (ED) and hospitalization rate, infection symptoms, new alloantibody formation, and antibiotic use during the 3-month study period. The investigators will compare groups using a Fisher exact test. Power: A difference of 20% will be of clinical interest. The investigators do not expect to have adequate power for this pilot study but at an alpha of 0.05 with 20 subjects in each group the investigators will be able to detect a difference of 47% between the proportions.
Time Frame: through fourth transfusion, an average of 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through study completion, a total of up to 24 weeks.
Arm/Group | ≤10 Day Blood | ≥30 Day Blood
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 3/13 | 5/13
Other Adverse Events (participants affected / at risk) | 4/13 | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ≤10 Day Blood (N=13) | ≥30 Day Blood (N=13)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Vaso-occlusive Pain (General disorders) | 2 (5) | 3 (4)
Acute Chest Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fistula Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ≤10 Day Blood (N=13) | ≥30 Day Blood (N=13)
Vaso-occlusive pain (General disorders) | 2 (2) | 4 (25)
Penile pain (General disorders) | 0 (0) | 1 (8)
Injury due to Fall (General disorders) | 1 (1) | 0 (0)
Fistula Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT03704922/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT03704922/ICF_000.pdf